CLINICAL TRIAL: NCT04031560
Title: Effects of an Integrative Program Combining Mindfulness-based Cognitive Therapy, Psychoeducation and Functional Remediation in Bipolar Disorder
Brief Title: Effects of an Integrative Psychological Program in Bipolar Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI17/00941
Record Dates: First submitted 2019-07-22; First posted 2019-07-24 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2023-08

CONDITIONS: Bipolar Disorder
Keywords: mindfulness; cognitive therapy; psychoeducation; functional remediation
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Integrative treatment
  Interventions: Behavioral: Integrative treatment
- Control (No Intervention): The control group (62 patients) will not receive any type of add-on psychotherapy.

INTERVENTIONS:
Behavioral: Integrative treatment — The experimental group (62 patients) will take part on the integrative group program consisting of 12-sessions, 90 minutes each, once a week (4 focused on psychoeducation, 1 directed to the family relatives, 3 on mindfulness and 4 on functional remediation)
  Arms: Experimental

SUMMARY:
Bipolar disorder is related to a high level of personal, familial, social and economic burden. There is a need for feasible adjunctive psychological interventions to use in clinical practice as a complement of pharmacotherapy to enhance aspects that medication cannot reach. This project aims at develop and evaluate the impact of an adjunctive brief integrative program for bipolar patients (euthymic or with subthreshold symptoms). The patients (N=124) will be randomly assigned to two different groups. The experimental group (62 patients) will take part on a group integrative program consisting of 12-sessions of 90 minutes (based on psychoeducation, mindfulness and functional remediation) whilst the control group (62 patients) will not receive any sort of add-on psychotherapy. All patients will mantain standard psychiatric treatment. Together with the baseline assessment, the whole sample will be assessed after the intervention and at 12 months from the baseline evaluation, regarding sociodemographic, clinical and neuropsychological variables. If the intervention is effective it will improve psychosocial functioning (main variable), wellbeing and quality of life, as well as improve clinical outcomes and neurocognitive functioning of those affected by the illness.

DETAILED DESCRIPTION:
Study design: Single-blind randomized control trial.

Participants: Study participants will be enrolled from the Bipolar Disorders Program of the Hospital Clinic of Barcelona (Spain) and the Bipolar Disorders Unit.

Procedure: At baseline, the sample will be evaluated with respect to sociodemographic, clinical and neuropsychological variables. Subsequently, patients will be randomly assigned (1:1) to two different groups. The experimental group (62 patients) will take part on the integrative group program consisting of 12-sessions, 90 minutes each, once a week (4 focused on psychoeducation, 1 directed to the family relatives, 3 on mindfulness and 4 on functional remediation) whilst the control group (62 patients) will not receive any type of add-on psychotherapy. All the patients will maintain a standard psychiatric treatment during the study. Together with the baseline assessment, the whole sample will be assessed after the intervention and at the 12 months of follow-up. Psychiatric medication will be recorded during the follow-up and the reasons for eventual modifications. All the subjects will be evaluated by researchers blinded to the treatment condition. Semi-structured interviews will be conducted and complemented with clinical records and with assessment instruments to collect variables related to the course of the illness. This study will be conducted in accordance with the ethical principles of the Declaration of Helsinki and Good Clinical Practice and approved by the Hospital Clinic Ethics and Research. All participants will be asked to provide written informed consent prior to their inclusion in the study.

Variables assessed:

1. Demographic variables: gender, age, marital status, educational status and work situation.
2. Clinical variables: age at the onset of BD, age at first hospitalization, total number and type of previous episodes, hospitalizations, history of psychotic symptoms, polarity of the first episode, seasonal pattern, presence of rapid cycling, bipolar subtype (I or II), comorbidities, familial psychiatric history, familial history of affective disorder, familial history of complete suicide, previous suicide attempts, number of attempts, method and medical severity of attempts, history of drug use.
3. Clinical scales: Temperament Evaluation of the Memphis, Pisa, Paris, and San Diego Autoquestionnaire (TEMPS-A, Akiskal et al, 2005), Barratts Impulsiveness Scale (BIS-11, Barratt et al, 1983), Biological Rhythms Interview of Assessment in Neuropsychiatry (BRIAN, Rosa et al., 2007), and Cognitive Complaints in Bipolar Disorder Rating Assessment (COBRA, Rosa et al., 2013).
4. Psychosocial functioning: Functional assessment short test (FAST, Rosa et al., 2007).
5. Wellbeing and quality of life: WHO (Five) Well Being Index (WHO, 1998), Quality of Life in Bipolar Disorder scale (QoL.BD, Michalak y Murray, 2010).
6. Scales of mindfulness: Five Facet Mindfulness Questionnaire (FFMQ, Baer et al., 2006), Mindful Attention Awareness Scale (MAAS, Brown y Ryan, 2003).
7. Neuropsychological assessment: WAIS-IV (Wechsler, 2012), with the following subtests: vocabulary, arithmetic, digit span, letter-number sequencing, symbol search, coding; Wisconsin Card Sorting Test (WCST, Heaton et al, 1981); Stroop Color-Word Interference Test (Golden y col., 1995); F-A-S Verbal Phonemic Fluency Test (Benton & Hamser, 1978); Trail Making Test (TMT, Reitan y Wolfson, 1985); Continuous Performance Test (CPT-III, Conners 2014); California Verbal Learning Test (CVLT-II, Delis et al, 2000); Rey-Osterrieth Complex Figure Test (Osterreith, 1944; Rey, 1941); the Mayer- Salovey-Caruso Emotional Intelligence Test (MSCEIT, Mayer et al., 2003) and the Iowa Gambling Test (IGT, Bechara et al, 1994).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of BD type I or II according to DSM-5 criteria
* euthymic or with subthreshold symptoms (HDRS <14; YMRS <8)
* absence of an acute mood episode in the 3 months prior to the beginning of the intervention

Exclusion Criteria:

* estimated Intelligence Quotient (IQ) lower than 85,
* significant physical or neurologic illness that can affect neuropsychological performance
* DSM-5 criteria of substance abuse or dependence
* inability to understand the purposes of the study
* absence of psychosocial interventions in the past 2 years (psychoeducation group, functional remediation, mindfulness)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 124 (Estimated)
Dates: Start 2018-03-25 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Psychosocial functioning measured by functioning assessment short test | 15 days
  The scale is interviewer-administered, designed for the assessment of psychosocial functioning. The 24 items of the scale are divided among 6 specific areas of functioning: autonomy, occupational functioning, cognitive functioning, financial issues, interpersonal relationships and leisure time. Each individual item is scored from 0 to 3. The global score (0-72) is obtained when the scores of each item are added up. The higher the score, the more serious the difficulties.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Sanchez-Moreno, Principal Investigator — Consorcio Centro de Investigación Biomédica en Red (CIBER)
Locations (1):
- Hospital Clinic of Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Valls E, Sanchez-Moreno J, Bonnin CM, Sole B, Prime-Tous M, Torres I, Brat M, Gavin P, Morilla I, Montejo L, Jimenez E, Varo C, Torrent C, Hidalgo-Mazzei D, Vieta E, Martinez-Aran A, Reinares M. Effects of an integrative approach to bipolar disorders combining psychoeducation, mindfulness-based cognitive therapy and functional remediation: Study protocol for a randomized controlled trial. Rev Psiquiatr Salud Ment (Engl Ed). 2020 Jul-Sep;13(3):165-173. doi: 10.1016/j.rpsm.2020.05.005. Epub 2020 Jul 7. English, Spanish. PMID 32651030
- [Result] Valls E, Bonnin CM, Torres I, Brat M, Prime-Tous M, Morilla I, Segu X, Sole B, Torrent C, Vieta E, Martinez-Aran A, Reinares M, Sanchez-Moreno J. Efficacy of an integrative approach for bipolar disorder: preliminary results from a randomized controlled trial. Psychol Med. 2021 Apr 16;52(16):1-12. doi: 10.1017/S0033291721001057. Online ahead of print. PMID 33858527